CLINICAL TRIAL: NCT05374629
Title: Exploring of the Effectiveness of the Shared-decision Making Education to the Patient With COPD: the Randomized-controlled Study
Brief Title: Study on the Effect of Smoking Cessation in COPD Patients After Shared Decision Making Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cathay General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CGH-109078
Record Dates: First submitted 2022-04-27; First posted 2022-05-16 (Actual); Last update posted 2022-05-16 (Actual); Status verified 2022-04

CONDITIONS: Copd; Smoking Cessation; Psychological Dependence
Keywords: COPD; shared decision making; smoking cessation; Psychological Cigarette Dependence
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Smoking Cessation

STUDY DESIGN:
Intervention Model Description: The intervention group had the shared decision-making of smoking cessation which was guided by the smoking cessation health educator. The control group received routine smoking cessation health education by another smoking cessation health educator. Both groups will receive a post-test three months after the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The Intervention group had Shared Decision Making of smoking cessation. (Experimental): The intervention group had the shared decision-making of smoking cessation which was guided by the smoking cessation health educator, and it containing the nicotine addiction, the impact of smoking on health, the methods and difficulties about smoking cessation, and the way of decision.
  Interventions: Behavioral: Use different methods of teaching
- The control group received routine smoking cessation health education (No Intervention): The control group received routine smoking cessation health education by another smoking cessation health educator, and it containing the harm of smoking, the benefits of quitting smoking, smoking cessation methods, and second-generation smoking cessation .

INTERVENTIONS:
Behavioral: Use different methods of teaching — Both groups will receive a smoking cessation education guideline and post-test three months after the intervention.
  Arms: The Intervention group had Shared Decision Making of smoking cessation.

SUMMARY:
There was no significant difference in the effectiveness of smoking cessation in COPD patients under a single session of SDM compared with a single session of smoking cessation education but significant improvement in the psychological dependence of smoking cessation shows that both groups. More intensive and more frequent interventions should be provided in the future.

DETAILED DESCRIPTION:
According to the World Health Organization (WHO), in 2016, 251 million people worldwide suffered from Chronic Obstructive Pulmonary Disease (COPD), accounting for 5% of the total number of global deaths, with an average of every 101 person dies from obstructive pulmonary disease in second. In 2020, the Taiwan Ministry of Health and Welfare's death cause statistics ranked COPD the eighth among the top ten causes of death in Taiwan, with 5,657 deaths. Among the main causes of death for people over 65 years old, it was found that COPD increases the risk with age. Since 2018, my country has It has entered an aging society since 2000, and the cause of death from chronic lower respiratory diseases aged 75-84 and over 85 has risen to the sixth and seventh respectively.

The purpose of this study is to explore the effect of shared decision-making services to the patients with COPD, and to understand the demographic variables, smoking-related variables, disease severity, and psychological dependence. The main purpose is to explore the association between the demographic variables of patients with COPD, smoking-related variables, disease severity variables including the severity of expiratory airflow obstruction, and the severity of the patient's current symptoms, and further analyze the differences of smoking cessation behavior and smoking psychological dependence index after giving smoking cessation Shared Decision Making.

The study involved a 3-months, single session intervention in a two-armed, randomized controlled trial, approved by the Institutional Review Board (IRB) of Cathay General Hospital (Taipei, Taiwan). Two groups of subjects participated: one with a Shared Decision Making smoking cessation intervention, and the other with usual care only.

A Chi-square test or t-test was employed to assess differences in sociodemographic variables, baseline physiological and biochemical detection and smoking behaviors. The paired t-test was used to assess the smoking cessation behavior, and examine variables related to smoking behavior with Pearson correlation. Finally, the linear regression was used to detected the association of smoking behavior with disease severity and smoking psychological dependence after adjusting for demographic variables.

All tests were analyzed at a 95% significance level (p<0.05). Intention-to-treat analysis was not used since the ethical policy stated that non-compliers who refused to continue to participate had to be excluded from the analysis. Analyses were conducted using PASW 22.0 software for windows (SPSS, Chicago, IL, USA).

ELIGIBILITY:
Inclusion Criteria:

* patients with COPD diagnosed by a physician.
* self-reported as a smoker
* 30 years old or above
* speak Chinese and Taiwanese
* agree to accept the questionnaire and inform consent.

Exclusion Criteria:

* Suffering from acute mental illness.
* Alcohol or other drug addicts.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2020-11-23 (Actual); Primary Completion 2022-02-10 (Actual); Study Completion 2022-02-10 (Actual)

PRIMARY OUTCOMES:
Smoking cessation success | 12weeks
  Ask smoking cessation behavior, answer success or failure by self.
Smoking cessation psychological dependence | 12weeks
  The smoking psychological dependence adopted the smoking psychological dependence scale proposed by ZL Huang and has obtained the authorization of the original author. It has a total of 37 questions, scale title including life connection and health concern, 1 point for strongly disagree, 2 points for disagree, 3 points for moderate, 4 points for agree, 5 points for strongly agree, plus total points. The minimum values is 37, maximum values is 185, the higher the score the more dependent it is. This scale has the internal consistency (Cronbach's alpha) of 0.94, and the two-week test-retest reliability was 0.77.

SECONDARY OUTCOMES:
The change of Fagerstrom Test for Nicotine Dependence (FTND) | baseline, pre-intervention
  Used the "Fagerstrom Test for Nicotine Dependence" (FTND) translated by Health Promotion Administration, Ministry of Health and Welfare. The content of the scale includes six questions. The total score is from 0 to 10, the higher the score, the higher the nicotine addiction, and it was divided into three categories: low addiction (0-3 points), moderate addiction (4-6 points), and high addiction (7-10 points).
Disease severity | baseline, pre-intervention
  Follow COPD treatment guidelines：The severity of expiratory airflow obstruction by the Forced expiratory volume in 1 second (FEV1) value, Mild ( FEV1 ≥ 80%), Moderate ( 50% ≤ FEV1 < 80%), Severe (30% ≤ FEV1 < 50%) and Extremely severe (FEV1 < 30%).

CONTACTS AND LOCATIONS:
Overall Officials: Yen-Ping Tsai, Principal Investigator — Cathay General Hospital
Locations (1):
- Cathay General Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Huang WH, Hsu HY, Chang BC, Chang FC. Factors Correlated with Success Rate of Outpatient Smoking Cessation Services in Taiwan. Int J Environ Res Public Health. 2018 Jun 10;15(6):1218. doi: 10.3390/ijerph15061218. PMID 29890766